CLINICAL TRIAL: NCT04310553
Title: An Open-label, Multicenter, Prospective Study of Irreversible Electroporation (Nano Knife) Combined With Radiotherapy and Chemotherapy in Patients With Locally Advanced Pancreatic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Ruijin Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPOG_006
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Pancreatic Cancer; Locally Advanced Pancreatic Caner
Keywords: irreversible electroporation, nano knife, pancreatic cancer.
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): This project plans to enroll 40 patients receiving nanoknife treatment, our center enrolls 20 patients, and the other two centers will enroll 10 patients each. The number of patients expected to participate in the study is 240.
  Interventions: Procedure: Irreversible electroporation

INTERVENTIONS:
Procedure: Irreversible electroporation — Patients with locally advanced pancreatic cancer diagnosed by cell / histopathology will receive nano knife treatment if the target lesion is not suitable for surgical resection or the target lesion is suitable for surgical resection but patients give up surgery and choose nano knife combined with chemotherapy. Patients who have not previously received first-line chemotherapy will receive systemic chemotherapy for 4-6 cycles of treatment. Imaging evaluation will be performed every 6-8 weeks (± 7 days) during chemotherapy.
  Other Names: Nano Knife

SUMMARY:
This is an open-label, multicenter, prospective study of irreversible electroporation (nano knife) combined with radiotherapy and chemotherapy in patients with locally advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, no gender limitation;
2. Patients with locally advanced pancreatic cancer diagnosed by cell / histopathology, either initially diagnosed or previously treated;
3. The target lesion is not suitable for surgical resection, or the target lesion is suitable for surgical resection but the patient gives up the surgical treatment and chooses nano-knife combined with radiotherapy and chemotherapy
4. ECOG score is 0 ~ 2;
5. Expected survival ≥ 3 months;
6. Women of childbearing age must undergo a pregnancy test within 14 days prior to enrollment, and those who have a negative result are eligible for enrollment. Men and women of childbearing age and their sexual partners agreed to use reliable methods of contraception before, during, and at least 90 days after the end of the study.
7. Full informed consent and signed informed consent.

Exclusion Criteria:

1. Patients suffering from active infection; high blood pressure (≥160 / 100mmHg) that cannot be controlled by drugs; angina pectoris and unstable angina pectoris that have begun in the last 3 months. Myocardial infarction and cardiac insufficiency occurred within 1 year before enrollment ≥ NYHA Class II), schizophrenia, or history of psychotropic substance abuse;
2. Patients with severe heart and lung insufficiency or intolerance to general anesthesia;
3. Those who are allergic to CT and MRI contrast agents and unable to perform preoperative three-phase dynamic enhanced scanning;
4. Ascites due to clinical symptoms, after 2 weeks of conservative medical treatment (excluding drainage of ascites), the ascites still increases gradually;
5. Pregnant or lactating women;
6. HBV DNA ≥ 104 copies or ≥ 2000 IU / mL, antiviral liver protection treatment is required before HBV-DNA <104 copies (2000 IU / mL) before enrollment, and continue to take antiviral drugs and monitor liver function And hepatitis B virus load; HCV antibody positive or HCV-RNA positive; HIV-infected patients;
7. Patients that the investigator considers unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | ±7 days
  according to RECIST1.1

SECONDARY OUTCOMES:
Time to progress | ±7 days
  according to RECIST1.1
progress free survival | ±7 days
  according to RECIST1.1
Observe response rate | ±7 days
  according to RECIST1.1
disease control rate | ±7 days
  according to RECIST1.1
clinical benefit rate, CBR | ±7 days
  EOLTC QLQ-C30 (V3.0 Chinese version) was used to evaluate the quality of life (QOL) according to the European Cancer Research and Treatment Organization (EORTC) core quality of life scale

CONTACTS AND LOCATIONS:
Overall Officials: Liwei Wang, MD, Principal Investigator — RenJi Hospital
Locations (1):
- RenJiH, Shanghai, Shanghai Municipality, China